CLINICAL TRIAL: NCT06259656
Title: Antibody Response to Coronavirus Disease 2019 (COVID-19) Vaccination in Pregnant Woman and Transplacental Passage Into Cord Blood.
Brief Title: Correlation of Antibody Response to COVID-19 Vaccination in Pregnant Woman and Transplacental Passage Into Cord Blood.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vachira Phuket Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VPH REC 009/2023
Record Dates: First submitted 2024-02-13; First posted 2024-02-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-10

CONDITIONS: Covid-19
Keywords: Anti SARs-CoV; Pregnancy; Cordblood; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Thai term pregnant women are recruited at labor room, after informed consent was done. Characteristic data (such as vaccination type and time) and Maternal Blood was collected then cord blood was collected after birth. All blood was sent to test Anti SARs CoV antibody level. Then all data and 80 test result will analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thai term pregnant woman who have at least One dose of Covid vaccination (Other): Maternal and cord blood was collected to test COVID-19 Spike Protein IgG Quantitative Antibody (CMIA)
  Interventions: Diagnostic Test: COVID-19 Spike Protein IgG Quantitative Antibody (CMIA)

INTERVENTIONS:
Diagnostic Test: COVID-19 Spike Protein IgG Quantitative Antibody (CMIA) — Maternal blood and cord blood were collected to test for COVID-19 Spike Protein IgG Quantitative Antibody (CMIA)

SUMMARY:
The goal of this study is to study the correlation of maternal and cord blood level of Anti SAR-CoV.

DETAILED DESCRIPTION:
The goal of this study is to study the correlation of maternal and cord blood level of Anti SAR-CoV. Sample size is 40 Thai patients at labor room Vachira Phuket Hospital in October - November 2023, who have at least one COVID-19 vaccination before or when pregnant. The Secondary outcome is to study time effect after COVID-19 vaccination and effect of vaccine type on Antibody level.

ELIGIBILITY:
Inclusion Criteria:

* Thai term pregnant women
* 18-45 year old
* At least 1 covid vaccination received
* admission at Vachira Phuket Hospital Labor Room

Exclusion Criteria:

* Do not want to participate
* Unstable or Emergency condition

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-25 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
COVID-19 Spike Protein IgG Quantitative Antibody (CMIA) Level | 1 month
  Test for correlation of level in maternal and cord blood

SECONDARY OUTCOMES:
Analysed time effect from last vaccination and type. | 1 month
  Test for time effect after last dose of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Vachira Phuket Hospital, Phuket, Thailand

IPD SHARING:
Plan to Share IPD: No